CLINICAL TRIAL: NCT00451932
Title: A Multicentre, Randomised, Double-Blind, Tacrolimus Dual Therapy-Controlled, Parallel Group, Multiple Oral Dose Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of FK778 in Liver Transplant Patients Receiving Standard Tacrolimus (FK506) and Steroids Therapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of FK778 in Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-778-01-100; 8778-CL-1200
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Liver Transplantation
Keywords: Malononitrilamide; Immunosuppression; treatment efficacy; treatment effectiveness
MeSH Terms: interventions — 2-cyano-3-hydroxy-N-(4-(trifluoromethyl)phenyl)-2-hepten-6-ynamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: FK778

SUMMARY:
A proof of concept study to evaluate the safety and effectiveness of FK778 in liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age and not older than 65 years.
* Female patients of child bearing potential must have a negative serum pregnancy test prior to enrollment and must agree to practice effective birth control during the study.
* Male patients must agree to practice effective birth control methods during the study.
* Patient is a recipient of a primary whole cadaveric liver transplant

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a liver.
* Patient has received an ABO incompatible donor liver.
* Patient or donor is known to be HIV positive.
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Patient is being transplanted for hepatic malignancy with a single nodule greater than 5.0 cm in diameter or 2 or more nodules with at least one > 3.0 cm.
* Patient has a serum creatinine >175 µmol/L at baseline. Patient has uncontrolled concomitant infections and/or severe diarrhoea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with the study objectives.
* Patient who is receiving or may require warfarin or fluvastatin during the study.
* Patient is participating in another clinical trial and/or is taking or has been taking an investigational drug in the 28 days prior to transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2002-10; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Event rate of biopsy-proven acute rejections

SECONDARY OUTCOMES:
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Universitätsklinik Charité
Locations (29):
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Leuven
- Canada (3):
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
- Czechia (2):
  - Brno
  - Prague
- France (6):
  - Clichy
  - Lyon
  - Montpellier
  - Rennes
  - Strasbourg
  - Villejuif
- Germany (4):
  - Berlin
  - Essen
  - Hamburg
  - Hanover
- Budapest, Hungary
- Italy (2):
  - Milan
  - Udine
- Rotterdam, Netherlands
- Spain (4):
  - Barakaldo
  - Barcelona
  - Madrid
  - Santiago de Compostela
- Zurich, Switzerland
- United Kingdom (2):
  - Birmingham
  - London